CLINICAL TRIAL: NCT00907270
Title: Effect of Vitamin D Supplementation on Leptin Resistance, Hunger, Body Weight and Resting Energy Expenditure in Obese Women.
Brief Title: Supplementation With Vitamin D Improves Leptin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mexican National Institute of Public Health (Other Government)
Responsible Party: Mario Flores-Aldana, National Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69770
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol: 400 IU/day (Active Comparator): Control: (n=50) Each subject will be evaluated after supplementation during six months with Vitamin D (Cholecalciferol: 400 IU/day)
  Interventions: Dietary Supplement: Cholecalciferol
- Cholecalciferol 4000 IU/day (Experimental): Experimental: (n=50) Each subject will be evaluated after supplementation during six months with Vitamin D
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Cholecalciferol: 4,000 IU/day and 400 IU/day
  Other Names: Cholecalciferol supplementation (400 IU and 4000 IU)

SUMMARY:
Participants will be randomly assigned in one of two groups. Group A: oral supplementation with 4,000 IU of vitamin D (cholecalciferol). Group B: oral supplementation with 400 IU of vitamin D (cholecalciferol). Both treatments will be consumed daily for 6 months.

Outcomes will be evaluated at baseline, three and six months. Variables related to leptin resistance will be evaluated.

The main hypothesis is that vitamin D will diminish leptin resistance in overweight and obese women. If the hypothesis is confirmed, women will show a reduction in the Resting energy expenditure: serum Leptin ratio (REE: Leptin ratio), as well as a reduction of hunger, body weight, body and abdominal fat and an increase in resting energy expenditure.

DETAILED DESCRIPTION:
Study subjects will get dietary advice and physical activity counseling. At the end of the study, participants with suboptimal vitamin D levels (<80 nmol/L 25-OH-D) will receive treatment to normalize their vitamin D status.

Variables related to leptin resistance like resting metabolic expenditure, hunger, body weight and human body fat will be assessed. Outcomes will include, glucose, insulin, C-reactive protein, inflammatory interleukins (IL-6 & TNF-α) and non-inflammatory interleukins (IL-10 & TGF-β-1).

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25-29.9
* Serum vitamin D levels: 20-80 nmol/L (25-OH-D)

Exclusion Criteria:

* Liver disease
* Kidney disease
* Diabetes mellitus
* Malignity
* Any kind of hormonal disorder
* Medication that modify hunger/satiety answer and those medications that alter -the glucose/insulin metabolism
* Subjects with diet treatment to lose weight

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of leptin resistance: (resting energy expenditure: leptin ratio) before and after (3 and 6 months) supplementation with vitamin D3 (cholecalciferol) 4,000 or 400 IU/day. | basal, third and sixth month

SECONDARY OUTCOMES:
Effect of vitamin D supplementation (25-OH-D): hunger, body weight, energy intake, resting energy expenditure, and body fat, improvement on low intensity chronic inflammation, SOCS-3 expression and JAK2/STAT3 signal. | Basal, third and sixth month

CONTACTS AND LOCATIONS:
Overall Officials: Mario Flores-Aldana, MsC, Principal Investigator — National Institute of public Health
Locations (1):
- National Institute of Social Insurance, Cuernavaca, Morelos, Mexico